CLINICAL TRIAL: NCT03405740
Title: Remote Patient Management of Cardiac Implantable Electronic Devices - Tachy
Brief Title: Remote Patient Management of CIEDs
Acronym: RPM CIED Tachy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ratika Parkash (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other); Abbott Medical Devices (Industry); Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Ratika Parkash, Staff Electrophysiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP005
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Patient Management (Active Comparator): Patients will be followed by remote monitoring only.
  Interventions: Device: Remote Patient Management
- Standard of Care (Placebo Comparator): Remote monitoring at 6 month intervals, alternating with yearly in-clinic visits at their usual site.
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Remote Patient Management — 1. Transmissions will occur at six monthly intervals, with no in-clinic visits. If there is an actionable event on the remote transmission, patients will be seen at their closest community clinic.
  2. All patients will be required to follow up with their family physician at least annually, and their cardiologist at least every 2 years.
  3. Patients will be contacted by phone at 6 months and 12 months to document their current health status (change in cardiovascular medications, any cardiovascular hospitalizations, in-clinic device checks, or any new cardiovascular testing completed since the last visit)
  4. VIRTUES access
  Arms: Remote Patient Management
Device: Standard of Care — No intervention
  Arms: Standard of Care

SUMMARY:
This is a Canadian multicenter randomized controlled trial to assess remote patient management. Patients will be randomized to remote patient management with VIRTUES versus usual care, and will be stratified by RemoteView vs no RemoteView utilization, as well as by center.

DETAILED DESCRIPTION:
Remote monitoring (RM) has been in use for over a decade and is now used in a blended system of in clinic visits and RM to provide CIED follow up. Prior studies have focused on this blended model of follow up. In this study, we propose a paradigm shift in CIED follow up care that is fully remote, supported by a patient-centered communication system permitting patients to have greater understanding of their CIED and its function. Patients would not have to leave their own communities to obtain state-of-the art care for their cardiac condition or their CIED. Given the burgeoning use of CIEDs (ICDs and PMs), the aging population and particularly in Canada where 19% of the inhabitants are in communities classified as 'rural', many have long distances to travel to reach a health care facility, it is of the utmost importance to take full advantage of available and developing technologies to improve CIED follow up beyond current recommendations. During the life of these patients, many issues may arise, such as atrial or ventricular arrhythmias that may result in syncope, stroke or sudden death, need for increased monitoring resulting from device advisories, or minor programming adjustments to improve device performance, or simply the need for enhanced surveillance as the device battery depletes and replacement is anticipated. New technology has become available that not only permits surveillance, but also permits communication back to the patient, and their respective providers regarding the status of these devices. The combination of technologies will result in a total care of CIEDs termed Remote Patient Management - CIED (RPM-CIED). The incorporation of enhanced monitoring capability, along with automatic recalibration of device settings, allows us to develop a new paradigm of remote patient management where after the patient receives their device, they would remain in the care of their local health team ('spokes') and no longer require travel to the specialized device clinics ('hubs') for follow-up. It creates capacity in the specialized centers to focus exclusively on the problematic cases by removing the need for routine checks.

There are two avenues of new technology that will be used in this study:

1. Remote View: this secure, web-based portal facilitates a virtual view of the device programming by the specialist in real-time while the patient is in their local clinic, thus avoiding patient travel to the specialized clinic (hub).
2. VIRTUES (Virtual Integrated Reliable Transformative User-driven E-health System): this portal has been developed by the Cardiac Arrhythmia Network of Canada to allow the patient to receive reports from the remote transmissions of their device.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a Medtronic, Abbott or Boston Scientific defibrillator/CRT-D capable of remote monitoring with Carelink, Merlin or Latitude.
2. Able to provide consent.
3. Age >/= 18 years

Exclusion Criteria:

1. No family physician or general practitioner
2. Inability to be referred to a specialist
3. Currently followed more than every 6 months by a Heart Function Clinic
4. Participation in another randomized clinical trial that impacts outcome
5. Unreliable automated capture verification by device in pacemaker dependent patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to major adverse cardiac event (primary safety outcome) | 18 months
  Time to a major adverse event, including: death, stroke, hospitalization for complications relating to the device system, cardiovascular hospitalization, syncope, device-related Emergency Department visits.
Time to a device-detected event (primary efficacy outcome) | 18 months
  The response time from a clinical event to a clinical decision in response to arrhythmias, cardiovascular disease progression, and device issues with remote patient management as compared to standard of care

SECONDARY OUTCOMES:
Medication Compliance | 18 Months
  Compliance will be measured according to current Canadian Cardiovascular Society Heart Failure Guidelines
Minimum programming compliance | 18 months
  Minimum ICD programming according to Canadian Heart Rhythm Society programming recommendations
Number of clinical events leading to a change in medication | 18 months
  Events detected by the ICD that lead to a clinical decision to change medication
Inappropriate ICD shocks | 18 months
  Number of inappropriate ICD shocks
Appropriate ICD shocks | 18 months
  Number of appropriate ICD shocks
Time to detection of ventricular arrhythmia events | 18 months
  device-detected ventricular fibrillation or ventricular tachycardia
Detection of atrial high-rate episodes | 18 months
  Device detected high-rate episodes greater than 6 minutes
Number of Cardiovascular-related ER visits | 18 months
  Number of cardiovascular-related visits (<24 hours)
Number of Device-Related ER visits | 18 Months
  ER visits (<24 hrs) for a device-related reason (including an audio signal from the device (beeping), shock(s), or a device complication requiring medical attention)
Rate of syncope | 18 months
  Syncope
Cost effectiveness | 18 months
  An economic evaluation will include a cost utility analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (12):
- Canada (12):
  - Foothills Hospital, Calgary, Alberta
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QEII HSC, Halifax, Nova Scotia
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Center, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital SacreCoeur, Montreal, Quebec
  - Hopital Laval, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No